CLINICAL TRIAL: NCT05964543
Title: A Phase I/II Clinical Trial to Evaluate the Safety Tolerance and Initial Efficacy of Q-1802 Combined With Standard Treatment in Patients With Gastrointestinal Tumors
Brief Title: The Safety and Efficacy of Q-1802 Combined With XELOX in Gastrointestinal Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: QureBio Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Q-1802-201
Record Dates: First submitted 2023-07-19; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Gastroesophageal Junction (GEJ) Adenocarcinoma
Keywords: Neoplasms
MeSH Terms: conditions — Adenocarcinoma; Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Intervention Model Description: Phase Ib: Dose escalation;Phase II:Arm A：Combined administration group Q-1802 plus XELOX,Arm B Standard treatment group: XELOX alone
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase Ib: Dose escalation Q-1802+XELOX, (Experimental): According to "3+3" design, a dose of Q-1802 with two dose groups from low to high and one cycle fixed-dose XELOX will be given in DLT observation period. After DLT observation period, Q-1802+XELOX will be given by investigator,s decision until the subject meets study treatment discontinuation criteria.
  Interventions: Drug: Q-1802 Injection,Oxaliplatin Injection,Capecitabine
- Phase II: Q-1802 + XELOX Vs XELOX ; (Placebo Comparator): Phase II:Participants will be randomized to group A and B. Group A:receive a dose of Q-1802 at Cycle 1 Day 1 followed by a same dose in subsequent cycles every 2 weeks. Additionally, participants will receive XELOX (capecitabine/oxaliplatin) treatment until investigator confirmed disease progression or a total of 8 treatments (each cycle is defined as approximately 21 days). Oxaliplatin is administered on day 1 of each cycle, whereas capecitabine is taken twice daily on days 1 through 14. After a maximum of 8 treatments of Oxaplatin, subjects may continue to receive Q-1802 a every 2 weeks each cycle and capecitabine every 3 weeks at the investigator's discretion until the subject meets study treatment discontinuation criteria. Group B:Participants will receive XELOX (capecitabine/oxaliplatin) treatment alone until a total of 8 treatments (each cycle is defined as approximately 21 days). subjects may continue to receive capecitabine every 3 weeks at the investigator's discretion.
  Interventions: Drug: Q-1802 Injection,Oxaliplatin Injection,Capecitabine

INTERVENTIONS:
Drug: Q-1802 Injection,Oxaliplatin Injection,Capecitabine — Q-1802：A dose Q-1802 will be administered intravenously Q2W. XELOX（oxaliplatin，capecitabin）: 21 days as a cycle Oxaliplatin will be administered 130mg/m2 as a 2-hour IV infusion,administer once on the first day, with 21 days as a cycle Capecitabine will be administered 1000mg/m2 orally twice daily (D1-D14),21ds is one cycle.
  Other Names: Q-1802,Oxaliplatin Injection,Xeloda

SUMMARY:
The main purpose of this study is to evaluate safety, tolerability and the efficacy of Q-1802 plus SOC compared with SOC. .Pharmacokinetics (PK) ,Pharmacodynamics (PD) of Q-1802 and the immunogenicity profile of Q-1802 will be evaluated as well.

DETAILED DESCRIPTION:
This study is a multicenter, open label, phase Ⅰb/Ⅱ clinical study conducted in unresectable patients with advanced or recurrent metastatic Claudin18.2 positive (medium and high expression) and HER-2 negative primary gastric adenocarcinoma or gastric esophageal junction adenocarcinoma. The Phase Ib dose escalation study included two dose groups each combined with the XELOX standard treatment regimen. Perform dose escalation to obtain MTD and/or RP2D doses for combined administration. The Phase II study adopted an open label parallel randomized controlled design. Further observe the efficacy and safety of Q-1802 combined with XELOX regimen in treating patients with moderate to high expression of Claudin 18.2, and compare and analyze the efficacy and safety of Q-1802 combined with XELOX regimen and XELOX regimen alone.

ELIGIBILITY:
Inclusion criteria：

Patients with at least one measurable lesion per RECIST (v1.1);

Patients with medium or high expression of Claudin18.2 in tumor tissue samples tested by immunohistochemistry in central laboratory were included;

Patients with untreated, unresectable advanced or metastatic gastric adenocarcinoma or gastroesophageal junction adenocarcinoma with negative HER-2 immunohistochemistry or FISH test (HER-2 immunohistochemistry 0/1+ confirmed by a qualified local or central laboratory, or 2+ confirmed negative by FISH test) were included;

Eastern Cooperative Oncology Group (ECOG) performance status score 0 or 1 at screening and no deterioration occurs within two weeks before enrollment;

Life expectancy period ≥ 12 weeks;

Patients who have sufficient baseline organ function.

Exclusion Criteria:

Receive anti-tumor treatment within 4 weeks before the first administration or within 5 half-lives of the treatment drug, whichever is shorter;

Patients who have previously used Claudin 18.2 products for treatment;

With uncontrolled diseases;

Who are allergic to the study drug or any of its components;

Patients with a history of other primary malignant tumors at the time of screening, except for cured skin Basal-cell carcinoma or Cutaneous squamous-cell carcinoma or cervical Carcinoma in situ.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events(TRAE) | From the first dose of study drug administration up to 30 days after the last study medication administration, up to 12months
  TRAE is defined as the AEs that the casual relationship of the AE is ralated to Q-1802
Objective response rate (ORR) | From the first dose of study drug administration up to 6 months after the last pts in,up to19 months
  ORR is defined as proportion of participants with complete response, partial response (CR+PR).

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From the first dose of study drug administration up to the last pts who disease progression or death which occurs first,up to 21months
  PFS is defined as the interval of time between the date of first treatment to the earliest date of disease progression or death which occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD, Principal Investigator — Department of Medical Oncology, Beijing
Locations (1):
- Beijing cancer hospical, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No